CLINICAL TRIAL: NCT01876251
Title: Phase 1b Study Of Docetaxel + Pf 03084014 In Metastatic Or Locally Recurrent/Advanced Triple Negative Breast Cancer
Brief Title: A Study Evaluating The PF-03084014 In Combination With Docetaxel In Patients With Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on June 24th, 2015 due to change in strategy of PF-03084014 development. There were no safety/efficacy concerns behind the decision.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A8641016; 2013-000659-41 (EudraCT Number)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer Metastatic
Keywords: Breast cancer metastatic; docetaxel; PF-03084014
MeSH Terms: interventions — nirogacestat; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-03084014 plus docetaxel (Experimental): PF 03084014 will be administered orally, continuously, twice daily at doses from 80 to 150 mg in combination with docetaxel given every 3 weeks at doses from 75 to 100 mg/m^2
  Interventions: Drug: PF-03084014; Drug: Docetaxel

INTERVENTIONS:
Drug: PF-03084014 — Tablet, 10 mg, twice a day
Drug: PF-03084014 — Tablet, 50 mg, twice a day
Drug: PF-03084014 — Tablet, 100 mg, twice a day
Drug: Docetaxel — Solution for IV infusion 75 mg/m^2, every 3 weeks
  Other Names: Taxotere
Drug: Docetaxel — Solution for IV infusion 100 mg/m^2, every 3 weeks

SUMMARY:
This study is aimed to determine the tolerability of the PF-03084014 plus docetaxel combination in patients with advanced breast cancer. Preliminary information about the efficacy of the combination will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer with evidence of a) metastatic or b) locally recurrent/advanced disease.

Exclusion Criteria:

* Prior treatment with a gamma secretase inhibitors or other Notch signaling inhibitors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2015-12-24 (Actual); Study Completion 2015-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, IDS Pharmacy, Birmingham, Alabama
  - Stanford Cancer Institute, Stanford, California
  - Stanford Hospital & Clinics-DRUG SHIPMENT ADDRESS only, Stanford, California
  - Stanford Hospital & Clinics, Stanford, California
  - Stanford Women's Cancer Center, Stanford, California
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute (KCI), Detroit, Michigan
  - UNC Cancer Hospital Infusion Pharmacy, Chapel Hill, North Carolina
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Belgium (2):
  - Jules Bordet Institut, Brussels
  - Grand Hopital de Charleroi, Charleroi
- Instituto Europeo di Oncologia, Milan, Italy
- Spain (2):
  - Instituto Catalan de Oncologia de L'Hospitalet de Llobregat(ICO), Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8641016&StudyName=A%20Study%20Evaluating%20The%20PF-03084014%20In%20Combination%20With%20Docetaxel%20In%20Patients%20With%20Advanced%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants were enrolled of whom 1 was not treated and therefore 29 participants are stated below as starting the study.
Groups:
- PF-03084014 100 mg BID + Docetaxel 75 mg/m^2: PF-03084014 100 milligrams (mg) was given orally via tablets twice daily (BID) in 21-day cycles. On Day 1 of each cycle, participants were administered docetaxel 75 mg/square meters (m^2) intravenously.
- PF-03084014 100 mg BID + Docetaxel 100 mg/m^2: PF-03084014 100 milligrams (mg) was given orally via tablets twice daily (BID) in 21-day cycles. On Day 1 of each cycle, participants were administered docetaxel 100 mg/square meters (m^2) intravenously.
- PF-03084014 150 mg BID + Docetaxel 75 mg/m^2: PF-03084014 150 milligrams (mg) was given orally via tablets twice daily (BID) in 21-day cycles. On Day 1 of each cycle, participants were administered docetaxel 75 mg/square meters (m^2) intravenously.
Period: Overall Study
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Started | 15 | 3 | 11
Completed | 0 | 0 | 0
Not Completed | 15 | 3 | 11
Not completed — Clinical progression | 1 | 0 | 0
Not completed — Death | 2 | 0 | 1
Not completed — Participant started new treatment | 1 | 0 | 1
Not completed — Participant refused further follow-up | 0 | 0 | 1
Not completed — Study terminated | 1 | 0 | 0
Not completed — Objective progression or relapse | 10 | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2 | Total
Number analyzed (Participants) | 15 | 3 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (13.9) | 43.3 (17.9) | 46.2 (12.6) | 49.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 11 | 29
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) in Cycle 1
Description: Any DLT event in Cycle 1: Grade 4 neutropenia lasting more than (>)7 days; febrile neutropenia (Grade more than or equal to [>=] 3 and body temperature >=38.5 degrees Celsius); Grade >=3 neutropenic infection; Grade >=3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia without bleeding; Grade >=3 toxicities (except those that had not been maximally treated); Grade 3 prolongation of time from electrocardiogram (ECG) Q wave to the end of the T wave corresponding to electrical systole (QT) corrected for heart rate (QTc) which persisted after correction of reversible causes; delay of 2 weeks in receiving next scheduled cycle due to persisting treatment-related toxicities; and failure to deliver at least 80% of planned dose during first cycle due to treatment-related toxicities.
Time Frame: Cycle 1 Days 1-21
Population: All enrolled participants who were eligible, received study treatment, and who either experienced DLT during the first cycle, or completed the 1-cycle observation period.
Measure: Number; unit: participants
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
participants | 1 | 1 | 4

2. Primary Outcome: Progression-free Survival (PFS) at 6 Months - Expansion Cohort
Description: The period from study entry until disease progression, death or date of last contact. Assessment of response was made using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Baseline till 6 months post-dose
Population: The 6-month PFS was evaluated only for the participants in the expansion cohort (PF-03084014 100 mg BID + docetaxel 75 mg/m^2). Due to early study termination, only 7 participants were treated in the expansion cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 7
months | 4.1 [1.3 to 8.1]

3. Secondary Outcome: Number of Participants With All Causality and Treatment-related Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Withdrawals Due to TEAEs
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent AEs (TEAEs) are defined as newly occurring AEs or those worsening after first dose. AEs comprised both SAEs and non-SAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Causality assessment was made by the investigator. Grading was per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) version 3.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening, Grade 5=death related to AE.
Time Frame: Baseline up to 28-35 days after treatment discontinuation (up to Day 280)
Population: All 29 participants who received study treatment were included in the AE summarization/analysis.
Measure: Number; unit: participants
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 15 | 3 | 11
participants
  All causality TEAEs | 15 | 3 | 11
  Treatment-related (TR) TEAEs | 15 | 3 | 11
  All causality SAEs | 4 | 3 | 6
  TR SAEs | 3 | 3 | 6
  Grade 3 or 4 TEAEs, all causality | 15 | 3 | 11
  Grade 3 or 4 TEAEs, TR | 15 | 3 | 11
  Grade 5 TEAEs, all causality | 1 | 0 | 1
  Grade 5 TEAEs, TR | 0 | 0 | 1
  Permanent withdrawal due to all causality TEAE(s) | 1 | 1 | 6
  Permanent withdrawal due to TR TEAE(s) | 1 | 1 | 4

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes, clinical chemistry, and urinalysis (dipstick).
Time Frame: Baseline up to 28-35 days after treatment discontinuation (up to Day 280)
Population: All 29 participants who received study treatment were included in the safety analyses.
Measure: Number; unit: participants
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 15 | 3 | 11
participants | 15 | 3 | 11

5. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: OR was based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 millimeters [mm]). No new lesions. PR was defined as more than or equal to (>=) 30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 6 weeks from Cycle 2 onwards up to 26 months
Population: All 29 participants who received study treatment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 15 | 3 | 11
percentage of participants | 13.3 [1.7 to 40.5] | 0 [0.0 to 70.8] | 18.2 [2.3 to 51.8]

6. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Time 0 to Time of Last Measured Concentration (AUClast) of PF-03084014 in Dose-finding Cohort
Description: Serum PF-03084014 pharmacokinetic (PK) parameters were calculated following twice daily (BID) doses of PF-03084014 given alone (Cycle 1 Day 21) and in combination with docetaxel (Cycle 1 Day 2 and Cycle 2 Day 1).
Time Frame: Cycle (C) 1 Days (D) 1, 2, 8, and 21; Day 1 of subsequent cycles and at EOT (max reached: Cycle 12)
Population: All 22 participants treated in the dose escalation stage were included in the analysis. n=number of evaluable participants at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)*hour (hr)/milliliter (mL)
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
nanogram (ng)*hour (hr)/milliliter (mL)
  C1D2 | 1779 (63) | 1380 (57) | 1839 (32)
  C1D21: number analyzed (Participants) | 7 | 3 | 8
  C1D21 | 4119 (39) | 3234 (21) | 5575 (59)
  C2D1: number analyzed (Participants) | 7 | 2 | 8
  C2D1 | 1983 (53) | NA (NA) — There were only 2 participants with reportable AUClast at this time point and summary statistics are not calculated for <3 participants. Individual values were 1350 and 1400 ng*hr/mL. | 2652 (28)

7. Secondary Outcome: AUClast and AUC From Time 0 Extrapolated to Infinite Time (AUCinf) of Docetaxel in Dose-finding Cohort
Description: Plasma docetaxel PK parameters were calculated following a 1-hr infusion of docetaxel given alone (Cycle 1 Day 1) and in combination with BID dosing of PF-03084014 (Cycle 2 Day 1)
Time Frame: C1D1, 2, 8, and 21; D1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)*hour (hr)/milliliter (mL)
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
nanogram (ng)*hour (hr)/milliliter (mL)
  AUClast, C1D1 | 3535 (113) | 4082 (36) | 2121 (49)
  AUClast, C2D1: number analyzed (Participants) | 7 | 2 | 8
  AUClast, C2D1 | 2377 (29) | NA (NA) — There were only 2 participants with reportable AUClast at this time point and summary statistics are not calculated for <3 participants. Individual values were 2270 and 1730 ng*hr/mL. | 2136 (47)
  AUCinf, C1D1: number analyzed (Participants) | 2 | 2 | 5
  AUCinf, C1D1 | NA (NA) — There were only 2 participants with reportable AUCinf at this time point and summary statistics are not calculated for <3 participants. Individual values were 30800 and 3020 ng*hr/mL. | NA (NA) — There were only 2 participants with reportable AUCinf at this time point and summary statistics are not calculated for <3 participants. Individual values were 2970 and 4490 ng*hr/mL. | 2509 (63)
  AUCinf, C2D1: number analyzed (Participants) | 6 | 1 | 3
  AUCinf, C2D1 | 2530 (30) | NA (NA) — There was only 1 participant with reportable AUCinf at this time point and summary statistics are not calculated for <3 participants. Individual value was 2410 ng*hr/mL. | 2929 (3)

8. Secondary Outcome: Maximum Serum or Plasma Concentration (Cmax) and Predose Concentration (Ctrough) of PF-03084014 in Dose-finding Cohort
Description: Serum PF-03084014 PK parameters were calculated following BID doses of PF-03084014 given alone (Cycle 1 Day 21) and in combination with docetaxel (Cycle 1 Day 2 and Cycle 2 Day 1)
Time Frame: C1D1, 2, 8, and 21; D1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
ng/mL
  Cmax, C1D2 | 884.8 (56) | 744.2 (51) | 896.6 (40)
  Cmax, C1D21: number analyzed (Participants) | 7 | 3 | 8
  Cmax, C1D21 | 1053 (51) | 677.5 (37) | 1501 (44)
  Ctrough, C1D21: number analyzed (Participants) | 7 | 3 | 8
  Ctrough, C1D21 | 214.7 (39) | 170.8 (36) | 306.1 (72)
  Cmax, C2D1: number analyzed (Participants) | 7 | 2 | 8
  Cmax, C2D1 | 885.7 (95) | NA (NA) — There were only 2 participants with reportable Cmax at this time point and summary statistics are not calculated for <3 participants. Individual values were 488 and 559 ng/mL. | 1100 (21)
  Ctrough, C2D1: number analyzed (Participants) | 7 | 2 | 8
  Ctrough, C2D1 | 186.1 (42) | NA (NA) — There were only 2 participants with reportable Ctrough at this time point and summary statistics are not calculated for <3 participants. Individual values were 116 and 129 ng/mL. | 226.4 (65)

9. Secondary Outcome: Cmax of Docetaxel in Dose-finding Cohort
Description: as for outcome 7
Time Frame: C1D1, 2, 8, and 21; D1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
ng/mL
  Cmax, C1D1 | 3711 (183) | 3447 (57) | 2103 (68)
  Cmax, C2D1: number analyzed (Participants) | 7 | 2 | 8
  Cmax, C2D1 | 2606 (29) | NA (NA) — There were only 2 participants with reportable Cmax at this time point and summary statistics are not calculated for <3 participants. Individual values were 2260 and 2200 ng/mL. | 1965 (35)

10. Secondary Outcome: Time to Cmax (Tmax) of PF-03084014 in Dose-finding Cohort
Description: as for outcome 8
Time Frame: C1D1, 2, 8, and 21; D1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
hr
  Tmax, C1D2 | 1.00 [0.500 to 1.03] | 1.02 [1.00 to 4.00] | 1.00 [0.500 to 1.03]
  Tmax, C1D21: number analyzed (Participants) | 7 | 3 | 8
  Tmax, C1D21 | 0.533 [0.417 to 1.00] | 1.00 [0.500 to 4.03] | 0.767 [0.500 to 2.00]
  Tmax, C2D1: number analyzed (Participants) | 7 | 2 | 8
  Tmax, C2D1 | 0.883 [0.000 to 1.00] | 1.03 [1.00 to 1.05] | 0.992 [0.500 to 1.02]

11. Secondary Outcome: Tmax of Docetaxel in Dose-finding Cohort
Description: as for outcome 7
Time Frame: C1D1, 2, 8, and 21; D1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
hr
  Tmax, C1D1 | 1.00 [0.500 to 1.05] | 0.917 [0.500 to 1.00] | 0.983 [0.500 to 1.05]
  Tmax, C2D1: number analyzed (Participants) | 7 | 2 | 8
  Tmax, C2D1 | 1.00 [0.517 to 1.03] | 0.767 [0.533 to 1.00] | 1.00 [0.500 to 1.50]

12. Secondary Outcome: Systemic Clearance (CL) of Docetaxel in Dose-finding Cohort
Description: as for outcome 7
Time Frame: C1D1, 2, 8, and 21; D1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)/hr
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
liter (L)/hr
  CL, C1D1: number analyzed (Participants) | 2 | 2 | 5
  CL, C1D1 | NA (NA) — There were only 2 participants with reportable CL at this time point and summary statistics are not calculated for <3 participants. Individual values were 5.59 and 41.8 L/hr. | NA (NA) — There were only 2 participants with reportable CL at this time point and summary statistics are not calculated for <3 participants. Individual values were 55.3 and 40.5 L/hr. | 55.51 (70)
  CL, C2D1: number analyzed (Participants) | 6 | 1 | 3
  CL, C2D1 | 51.97 (23) | NA (NA) — There was only 1 participant with reportable CL at this time point and summary statistics are not calculated for <3 participants. Individual value was 68.1 L/hr. | 45.40 (5)

13. Secondary Outcome: Terminal Half-life (t1/2) of Docetaxel in Dose-finding Cohort
Description: as for outcome 7
Time Frame: C1D1, 2, 8, and 21; D1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
hr
  t1/2, C1D1: number analyzed (Participants) | 2 | 2 | 5
  t1/2, C1D1 | 18.35 (NA) — There were only 2 participants with reportable t1/2 at this time point so standard deviation is not calculated for. Individual values were 20.8 and 15.9 hrs. | 6.555 (NA) — There were only 2 participants with reportable t1/2 at this time point so standard deviation is not calculated for. Individual values were 10.1 and 3.01 hrs. | 7.624 (5.368)
  t1/2, C2D1: number analyzed (Participants) | 6 | 1 | 3
  t1/2, C2D1 | 5.500 (7.259) | NA (NA) — There was only 1 participant with reportable t1/2 at this time point and summary statistics are not calculated for <3 participants. Individual value was 3.84 hr. | 14.27 (3.420)

14. Secondary Outcome: Volume of Distribution (Vss) of Docetaxel in Dose-finding Cohort
Description: as for outcome 7
Time Frame: C1D1, 2, 8, and 21; D1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 8 | 3 | 11
L
  Vss, C1D1: number analyzed (Participants) | 2 | 2 | 5
  Vss, C1D1 | NA (NA) — There were only 2 participants with reportable Vss at this time point and summary statistics are not calculated for <3 participants. Individual values were 5.54 and 288 L. | NA (NA) — There were only 2 participants with reportable Vss at this time point and summary statistics are not calculated for <3 participants. Individual values were 301 and 27.8 L. | 97.34 (73)
  Vss, C2D1: number analyzed (Participants) | 6 | 1 | 3
  Vss, C2D1 | 57.37 (127) | NA (NA) — There was only 1 participant with reportable Vss at this time point and summary statistics are not calculated for <3 participants. Individual value was 85.4 L. | 231.5 (25)

15. Secondary Outcome: AUClast of PF-03084014 in the Expansion Cohort
Time Frame: C1D1, C1D21, and Day 1 of subsequent cycles and at EOT (max reached: C12)
Population: All 7 participants who received treatment in the expansion cohort were included in the analysis. n=number of evaluable participants at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 7
ng*hr/mL
  AUClast, C1D1 | 1098 (47)
  AUClast, C1D21: number analyzed (Participants) | 5
  AUClast, C1D21 | 1955 (16)

16. Secondary Outcome: Cmax of PF-03084014 in the Expansion Cohort
Time Frame: C1D1, C1D21, and Day 1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 7
ng/mL
  Cmax, C1D1 | 496.7 (70)
  Cmax, C1D21: number analyzed (Participants) | 5
  Cmax, C1D21 | 982.1 (20)

17. Secondary Outcome: Tmax of PF-03084014 in the Expansion Cohort
Time Frame: C1D1, C1D21, and Day 1 of subsequent cycles and at EOT (max reached: C12)
Population: as for outcome 15
Measure: Median (Full Range); unit: hr
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 7
hr
  Tmax, C1D1 | 0.983 [0.500 to 1.00]
  Tmax, C1D21: number analyzed (Participants) | 5
  Tmax, C1D21 | 1.00 [0.483 to 1.00]

18. Secondary Outcome: Ctrough of PF-03084014 in the Expansion Cohort
Time Frame: C1D1, C1D21, and Day 1 of subsequent cycles and at EOT (max reached: C12)
Population: All 7 participants who received treatment in the expansion cohort were included in the analysis. At Cycle 1 Day 21, only 5 participants had available data for Ctrough.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 5
ng/mL | 89.22 (51) [0.500 to 1.00]

19. Secondary Outcome: Duration of Response (DR)
Description: Duration of response (DR) defined as time from start of first documented objective tumor response [Complete Response (CR) or Partial Response (PR)] to first documented objective tumor progression or death due to any cause, whichever occurs first. DR = (the end date for DR minus first subsequent confirmed CR or PR plus 1) divided by 7.02. CR: disappearance of all target lesions. PR: at least 30% decrease in the sum of diameters of target lesions.
Time Frame: Baseline up to 28-35 days after treatment discontinuation (up to Day 280)
Population: Only 4 participants had CR or PR, 2 each in the PF-03084014 100 mg BID + docetaxel 75 mg/m^2 and PF-03084014 150 mg BID + docetaxel 75 mg/m^2 groups.
Measure: Number; unit: months
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 2 | 2
months | NA — Summary statistics not provided as there were 2 participants with PR/CR. Individual DRs were 2.79 and 5.55 months. | NA — Summary statistics not provided as there were 2 participants with PR/CR. Individual DRs were 3.19 and 4.20 months.

20. Secondary Outcome: Number of Participants With QTc Values Meeting Categorical Summarization Criteria
Description: Criteria for categorical summarization of the time corresponding to the beginning of depolarization to repolarization of the ventricles (QT) corrected for heart rate (QTc) using Bazett's correction (QTcB) or Fridericia's correction (QTcF) included: maximum QTcB or QTcF less than or equal to (<=) 450 milliseconds (msec), 450 to <=480 msec, 480 to <=500 msec, more than (>) 500 msec; maximum QTcB or QTcF changes (increases/decreases) from baseline (BL) less than (<) 30 msec, 30 to <60 msec, more than or equal to (>=) 60 msec.
Time Frame: Screening, C1D1, C1D21, Day 1 of subsequent cycles, and EOT (maximum reached: C12)
Population: All 29 participants who received study treatment were analyzed for safety.
Measure: Number; unit: participants
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 15 | 3 | 11
participants
  QTcB <=450 msec | 7 | 1 | 2
  QTcB 450 to <=480 msec | 6 | 1 | 8
  QTcB 480 to <=500 msec | 2 | 1 | 1
  QTcB >500 msec | 0 | 0 | 0
  QTcF <=450 msec | 13 | 2 | 6
  QTcF 450 to <=480 msec | 1 | 0 | 5
  QTcF 480 to <=500 msec | 1 | 1 | 0
  QTcF >500 msec | 0 | 0 | 0
  QTcB increase from BL <30 msec | 11 | 3 | 6
  QTcB increase from BL 30-<60 msec | 4 | 0 | 5
  QTcB increase from BL >=60 msec | 0 | 0 | 0
  QTcF increase from BL <30 msec | 14 | 3 | 9
  QTcF increase from BL 30-<60 msec | 1 | 0 | 2
  QTcF increase from BL >=60 msec | 0 | 0 | 0
  QTcB decrease from BL <30 msec | 15 | 3 | 11
  QTcB decrease from BL 30-<60 msec | 0 | 0 | 0
  QTcB decrease from BL >=60msec | 0 | 0 | 0
  QTcF decrease from BL <30 msec | 13 | 3 | 8
  QTcF decrease from BL 30-<60 msec | 2 | 0 | 3
  QTcF decrease from BL >=60 msec | 0 | 0 | 0

21. Secondary Outcome: Percentage Change From Baseline in Notch 1 to 4 Ribonucleic Acid (RNA) in Blood
Description: As PF-03084014 acts on the Notch pathway as an inhibitor, it is of interest to investigate its effects, if any, on the Notch family of receptors, mainly Notch 1-4.
Time Frame: C1D1, C1D2, C1D8, C1D21 and EOT (maximum reached: C12)
Population: All treated participants who had at least 1 screening and post treatment biomarker assessment. n=number of evaluable participants for the specified biomarker at the specified time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Number analyzed (Participants) | 7 | 2 | 10
percentage change
  Notch 1 RNA, C1D1 | 4.240 (0.5164) | 3.990 (0.4581) | 4.431 (1.1781)
  Notch 1 RNA, C1D2 | -5.797 (11.0169) | -7.358 (14.6569) | -10.647 (19.1488)
  Notch 1 RNA, C1D8: number analyzed (Participants) | 7 | 1 | 9
  Notch 1 RNA, C1D8 | 32.557 (22.0342) | 60.199 (NA) — Only 1 participant was evaluable at this time point. | 35.305 (19.4523)
  Notch 1 RNA, C1D21: number analyzed (Participants) | 5 | 2 | 7
  Notch 1 RNA, C1D21 | 6.118 (17.0382) | 17.047 (15.6705) | 11.214 (7.9496)
  Notch 1 RNA, EOT: number analyzed (Participants) | 7 | 2 | 8
  Notch 1 RNA, EOT | 5.653 (12.0722) | 18.066 (9.4153) | 4.177 (14.6678)
  Notch 2 RNA, C1D1 | 4.139 (0.4344) | 3.856 (0.8869) | 4.351 (0.7672)
  Notch 2 RNA, C1D2 | -12.830 (8.1864) | -9.617 (16.7632) | -15.441 (20.3566)
  Notch 2 RNA, C1D8: number analyzed (Participants) | 7 | 1 | 9
  Notch 2 RNA, C1D8 | 15.426 (22.0876) | 43.069 (NA) — Only 1 participant was evaluable at this time point. | 17.234 (18.0896)
  Notch 2 RNA, C1D21: number analyzed (Participants) | 5 | 2 | 7
  Notch 2 RNA, C1D21 | 2.161 (9.7434) | 9.756 (22.6330) | 4.985 (7.6829)
  Notch 2 RNA, EOT: number analyzed (Participants) | 7 | 2 | 8
  Notch 2 RNA, EOT | -1.250 (11.6223) | 9.478 (28.0500) | -1.558 (10.9137)
  Notch 3 RNA, C1D1: number analyzed (Participants) | 1 | 1 | 5
  Notch 3 RNA, C1D1 | 14.250 (NA) — Only 1 participant was evaluable at this time point. | 14.673 (NA) — Only 1 participant was evaluable at this time point. | 14.765 (1.3469)
  Notch 3 RNA, C1D2: number analyzed (Participants) | 0 | 1 | 3
  Notch 3 RNA, C1D2 |  | 0.311 (NA) — Only 1 participant was evaluable at this time point. | -1.186 (2.9388)
  Notch 3 RNA, C1D8: number analyzed (Participants) | 1 | 1 | 4
  Notch 3 RNA, C1D8 | -2.532 (NA) — Only 1 participant was evaluable at this time point. | 4.608 (NA) — Only 1 participant was evaluable at this time point. | -0.154 (11.1968)
  Notch 3 RNA, C1D21: number analyzed (Participants) | 0 | 1 | 2
  Notch 3 RNA, C1D21 |  | 1.362 (NA) — Only 1 participant was evaluable at this time point. | -11.274 (19.4623)
  Notch 4 RNA, C1D1: number analyzed (Participants) | 4 | 1 | 6
  Notch 4 RNA, C1D1 | 13.903 (0.5575) | 13.228 (NA) — Only 1 participant was evaluable at this time point. | 14.309 (1.3340)
  Notch 4 RNA, C1D2: number analyzed (Participants) | 0 | 1 | 3
  Notch 4 RNA, C1D2 |  | 12.215 (NA) — Only 1 participant was evaluable at this time point. | 2.484 (5.9621)
  Notch 4 RNA, C1D8: number analyzed (Participants) | 2 | 0 | 6
  Notch 4 RNA, C1D8 | -13.264 (3.5374) |  | -9.427 (9.8077)
  Notch 4 RNA, C1D21: number analyzed (Participants) | 1 | 1 | 3
  Notch 4 RNA, C1D21 | 0.927 (NA) — Only 1 participant was evaluable at this time point. | 5.616 (NA) — Only 1 participant was evaluable at this time point. | -0.500 (6.4382)
  Notch 4 RNA, EOT: number analyzed (Participants) | 2 | 1 | 5
  Notch 4 RNA, EOT | -3.634 (9.0629) | 11.821 (NA) — Only 1 participant was evaluable at this time point. | -9.975 (9.8833)

ADVERSE EVENTS:
Time Frame: Baseline up to 28-35 days after treatment discontinuation (up to Day 280)
Description: All treated participants were analyzed for AEs. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2
Serious Adverse Events (participants affected / at risk) | 4/15 | 3/3 | 6/11
Other Adverse Events (participants affected / at risk) | 15/15 | 3/3 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 (N=15) | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 (N=3) | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2 (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03084014 100 mg BID + Docetaxel 75 mg/m^2 (N=15) | PF-03084014 100 mg BID + Docetaxel 100 mg/m^2 (N=3) | PF-03084014 150 mg BID + Docetaxel 75 mg/m^2 (N=11)
Anaemia (Blood and lymphatic system disorders) | 10 | 1 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 10 | 2 | 5
Neutropenia (Blood and lymphatic system disorders) | 12 | 3 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Diplopia (Eye disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 6 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 10 | 2 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 3 | 8
Oedema mouth (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 4
Vomiting (Gastrointestinal disorders) | 5 | 1 | 9
Asthenia (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 12 | 2 | 11
Influenza like illness (General disorders) | 1 | 0 | 2
Local swelling (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 9 | 2 | 3
Oedema peripheral (General disorders) | 3 | 1 | 1
Pain (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 3 | 4
Vessel puncture site bruise (General disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Candida infection (Infections and infestations) | 2 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 2
Pulpitis dental (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 2 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 1
Eosinophil count decreased (Investigations) | 0 | 0 | 1
International normalized ratio increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Monocyte count decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 1 | 1 | 1
White blood cell count decreased (Investigations) | 2 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 2 | 3
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 4 | 2 | 6
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 4 | 1 | 2
Breast inflammation (Reproductive system and breast disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 1
Vulvovaginal rash (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 2 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 6
Rash erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.